CLINICAL TRIAL: NCT04474600
Title: The Influence of Type of Anesthesia on Postoperative Renal Function After Nephrectomy: a Randomized Controlled Study
Brief Title: Anesthesia and Acute Kidney Injury After Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Kyu Yoon, clinical assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Anesthetics_Nx_AKI
Record Dates: First submitted 2020-07-07; First posted 2020-07-17 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Nephrectomy
Keywords: Anesthesia; Propofol; Inhaled anesthetics; Acute kidney injury; Nephrectomy
MeSH Terms: conditions — Acute Kidney Injury | interventions — Propofol; Desflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TIVA group (Experimental): Patients receiving the total intravenous anesthesia using propofol
  Interventions: Drug: Propofol
- Inhalation group (Active Comparator): Patients receiving inhalation anesthesia using desflurane
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Propofol — The induction and maintenance of anesthesia was performed by total intravenous anesthesia using propofol. In both groups, remifentanil is continuously infused throughout the surgery.
  Arms: TIVA group
Drug: Desflurane — The induction and maintenance of anesthesia was performed by inhalation anesthesia using desflurane. In both groups, remifentanil is continuously infused throughout the surgery.
  Arms: Inhalation group

SUMMARY:
This study investigates the influence of type of anesthesia on postoperative renal dysfunction in patients undergoing nephrectomy. The participants will be allocated to either the group receiving the total intravenous anesthesia (TIVA) using propofol or the group receiving the inhaled anesthetics using desflurane.

DETAILED DESCRIPTION:
Nephrectomy is considered as a standard therapy for renal cell carcinoma, but it can cause postoperative renal dysfunction, such as acute kidney injury and chronic kidney disease. Therefore, it is imperative to identify modifiable risk factors for postoperative acute kidney injury after nephrectomy in advance. According to a recent retrospective study, total intravenous anesthesia using propofol is significantly associated with lower incidence of acute kidney injury after nephrectomy, compared to the inhalation anesthesia. However, there is no prospective study which investigates the influence of type of anesthesia on postoperative renal function after nephrectomy. Therefore, in the present study, we aimed to investigate the influence of type of anesthesia on acute kidney injury after nephrectomy by performing randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients scheduled for elective open nephrectomy

Exclusion Criteria:

* Patients diagnosed with acute kidney injury preoperatively
* Patients who have chronic kidney disease over stage 5 (estimated glomerular filtration rate [eGFR] <15 ml/kg/1.73m2) or have regular hemodialysis preoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
the incidence of acute kidney injury | during the postoperative seven days
  acute kidney injury (diagnosed by KDIGO criteria)

SECONDARY OUTCOMES:
serum creatinine | postoperative day 1, 3, 14
  postoperative result of serum creatinine
estimated glomerular filtration rate | postoperative day 1, 3, 14
  postoperative result of estimated glomerular filtration rate
biomarker of renal injury | postoperative day 1, 3, 14
  postoperative result of biomarker of renal injury
the incidence of postoperative complications | during the postoperative two weeks
  urine leakage, prolonged ileus, wound infection, retroperitoneal abscess, pneumonia, reoperation, etc.
Length of hospital stay | during the postoperative two weeks
  length of hospital stay
Length of intensive care unit stay | during the postoperative two weeks
  length of intensive care unit stay

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No